CLINICAL TRIAL: NCT07284147
Title: Clinical Study on the Control Effect of 3D Designed Defocus Lenses on Myopia in Children and Adolescents
Brief Title: 3D Designed Defocus Lenses on Myopia Control in Children and Adolescents
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QX-2025-A-012
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Myopia Progressing
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 3D lens (Experimental): 3D Designed Defocus Lenses
  Interventions: Device: Defocus Lenses
- Control: H. A. L. T, highly aspheric lenslet technology (Active Comparator): H. A. L. T, highly aspheric lenslet technology
  Interventions: Device: Defocus Lenses

INTERVENTIONS:
Device: Defocus Lenses — Defocus Lenses on Myopia Control

SUMMARY:
This study aims to evaluate the effectiveness of lenses with 3D Designed Defocus in controlling the progression of myopia in children and adolescents, and to explore the feasibility of effective design, and apply personalized frame lenses for myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

Age: 6-14 years old; After using 1% cyclohexanone hydrochloride eye drops (Saifeijie) for ciliary muscle paralysis, binocular spherical power were within -0.40D~-4.00D, binocular cylinder power ≤ 1.50D, the anisometropia is ≤ 1.50D, the progression of myopia in the past year is greater than 0.5D, the best corrected far vision is at least 4.8, and the near vision is at least 5.0; Within 3 months, the myopia prevention and control methods such as multifocal glasses, orthokeratology, defocusing flexible glasses, progressive glasses, atropine eye drops, red light and acupuncture and moxibustion treatment were not used; The subject has a willingness to receive treatment and an informed consent form is signed by their legal guardian.

Exclusion Criteria:

-

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Subjective refraction equivalent spherical | 12 months
  Subjective refraction equivalent spherical

SECONDARY OUTCOMES:
Axial length | 12 months
  Axial length
Choroidal thickness | 12 months
  Choroidal thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Diseases Prevention &Treatment Center/ Shanghai Eye Hospital, School of Medicine, Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided